CLINICAL TRIAL: NCT04497753
Title: An Epidemiological Investigation on Correct Wearing of Mask by Hood Test
Status: Completed | Type: Observational
Sponsor: Fuwai Yunnan Cardiovascular Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-KZLXB-02-02
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Respiratory Infectious Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Can't fell bitterness: 1. The subject wears a mask and a hood, opens his/her mouth to breathe, and sticks out his/her tongue properly. Using the fitness test reagent to spray into the hood, the number of sprays should be the same as that of the sensitivity test.
  2. Record whether the subject feels bitterness, if there is no feeling, the test is over.
- Can fell bitterness: 1. The subject wears a mask and a hood, opens his/her mouth to breathe, and sticks out his/her tongue properly. Using the fitness test reagent to spray into the hood, the number of sprays should be the same as that of the sensitivity test.
  2. Record whether the subject feels bitterness, If there is a sensation, put the adhesive strip on the upper edge of the subject's mask and put on the hood to carry out the above fitness test again.
  3. Record whether the subject feels bitterness, if not, the test is over. If there is any sensation, ask the subject to change to a medical surgical mask, and put an adhesive strip on the upper edge of the mask, and put on the hood to carry out the above fitness test again.

SUMMARY:
The purpose of this study was to explore the relationship between the transmission of respiratory diseases and the correct wearing of masks, as well as the factors affecting the correct wearing of masks. The research is beneficial to the prevention of respiratory diseases and moves the barrier of prevention and control forward. It is of great significance to COVID-19 's practical prevention and control.

DETAILED DESCRIPTION:
1. Overall design：This study uses the methods of cross-sectional survey and chance sampling.
2. Sign the Informed Consent Form.
3. Investigation on the basic situation of personnel: The gender, age and education level of the subjects were analyzed as the factors influencing whether the mask was worn correctly or not.
4. Investigation on the types of wearing masks： 1) The types of masks worn by the subjects were recorded as the basis of stratified statistics.

2) Mask suitability testing：

1. Visual inspection whether the mask is close to the face with obvious gaps.
2. Breathing test Are there any obvious gaps or whether the cotton around the mask is blown when the subject taking a deep breath.
3. Spray test The FT-30 qualitative fitness test system of 3M company was used to test the suitability and correctness of wearing mask.

In the spray test, all subjects underwent a sensitivity test to prove their ability to smell the bitterness of the reagent, and then sensitive subjects can participate in the hood test..

In order to objectively reflect the overall situation of the subjects, it is necessary to cover many ages and educational levels of men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy people with autonomous behavior ability and language expression ability who are older than or equal to 7 years old, Persons under the age of 18 need to obtain the consent of their legal guardians；
2. The subjects and / or their legal guardians have the ability to understand the contents of the study and to participate in all the research processes with the subjects；
3. People who volunteered to take part in the study；
4. There was no respiratory infection in nearly one month.

Exclusion Criteria:

1. People with a history of allergies, including those who are allergic to pollen, dust mites, etc；
2. People with any history of drug allergy；
3. People who have participated in the experiment are not allowed to participate in this study for the second time;
4. Pregnant women；
5. The healer after COVID-19 's infection；
6. After questioning, it was found that the subjects were the factors that affected the study, such as dysosmia, or those who had decreased olfactory ability due to disease, or facial paralysis, which affected the judgment of the test；
7. Those who are participating in clinical trials of other drugs / devices；
8. Subjects with poor compliance or unwilling to cooperate with the operation as required；
9. The researchers believe that any other situation that may affect the evaluation of the study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Those who are 7 years old or above, have the ability of autonomous behavior and language expression, are willing to take the test.
Sampling Method: Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
can or can't fell bitterness | Immediately after spray test
  Whenever the subject feels bitter, it means that the mask does not fit well with the subject's face.
  If the subjects do not feel bitter all the time, it means that the mask is suitable for the subjects' face and can be worn.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Duo, Principal Investigator — Fuwai Yunnan Cardiovascular Hospital
Locations (8):
- China (8):
  - Fuwai hospital, Beijing, Beijing, Beijing Municipality
  - Taizhou Health Bureau, Taizhou, Jiangsu
  - Bin Health Wen, Jinzhong, Shanxi
  - Yuanqu Health Bureau, Yuncheng, Shanxi
  - Fuwai Yunnan Cardiovascular Hospital, Kunming, Yunnan
  - Luliang Health Bureau, Qujing, Yunnan
  - Shizong Health Bureau, Qujing, Yunnan
  - Luoping Health Bureau, Qujing, Yunnan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT04497753/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT04497753/Prot_SAP_003.pdf